CLINICAL TRIAL: NCT00763724
Title: A Propensity-Matched Retrospective Cohort Study of Antidepressant Drug Exposure and Risk of Suicide Attempt in Adults From a Large U.S. Managed Care Population
Brief Title: Antidepressant Drug Exposure and Risk of Suicide Attempt Resulting in Medical Intervention in US Adults
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 12016; F1J-MC-B027
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Depression; Suicide
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 1: Duloxetine
- 2: Venlafaxine
- 3: SSRI
- 4: TCA
- 5: Multiple Antidepressants
- 6: Depressed (not antidepressant treated)
- 7: General population

SUMMARY:
The primary objective of the study is to estimate the incidence of suicide attempts resulting in a medical encounter or hospitalization in seven propensity matched cohorts of subjects: patients treated with duloxetine for depression, patients treated with one of three other antidepressants or antidepressant classes (venlafaxine, SSRIs, or TCAs) for depression, patients treated with multiple antidepressants for depression (either concurrently or consecutively), depressed patients with no pharmacologic treatment, and a non-depressed general population sample.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at index date
* Have at least 6 months of continuous enrollment data prior to index date.
* Have complete medical, facility, and pharmacy records (the latter of which will include complete quantity and days supplied information).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be based on data from the PharMetrics Patient-Centric Database, a commercially available claims database provided by PharMetrics, Inc., a Unit of IMS.
Sampling Method: Non-Probability Sample
Enrollment: 254432 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence of suicide attempt resulting in medical encounter or hospitalization. | Endpoint

SECONDARY OUTCOMES:
Relative risk of suicide attempt resulting in medical encounters or hospitalization | Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon-Fri 9am - 5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company